CLINICAL TRIAL: NCT05180123
Title: Clinical and MRI Evaluation of ACL Reconstruction Results in Adolescents With Follow-up at Least 3 Years.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMMHRI-BCO.37/2019-A
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: ACL Injuries; Knee Instability
Keywords: Anterior cruciate ligament; ACL; Knee injuries; Adolescents; ACL injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients after ACL reconstruction in adolescence (Other)
  Interventions: Procedure: Anterior cruciate ligament reconstruction

INTERVENTIONS:
Procedure: Anterior cruciate ligament reconstruction — Adolescent patients with confirmed full thickness ACL injury were operated arthroscopically with semitendinosus and gracilis autograft anatomical reconstruction.

SUMMARY:
In this retrospective research results of ACL reconstruction in adolescent will be evaluated. As we know ACL ruptures become more frequent and more often operated these days. According to literature the results in patients younger than 20 years old are worse. Therefore clinical and MRI evaluation will be performed. The aim of the study is to assess subjective and objective functional outcome of ACL reconstruction with follow-up at least 3 years. MRI scans will be evaluated to highlight any early signs of osteoarthritis and describe graft morphology. IKDC, KOOS scales will be utilised for subjective evaluation. Clinical tests such as Lachman's, pivot shift, Appley's along with anterior tibial shift measurement with digital arthrometer for objective assessment will be also performed. Additionally isokinetic tests will be performed in two speeds of 60 and 180 deg/s. Most of important isokinetic parameters such as peak torque, torque in 30 deg, time to peak torque, peak torque to body weight both for quadriceps and hamstrings will be measured .

Preliminary group of patients consists of 150 cases with follow-up at least 3 years, operated in age 12-17 years. All cases available for the study will be assessed with methodology above. Dedicated statistical test will be utilised to evaluate the results.

ELIGIBILITY:
Inclusion Criteria:

* age between 10-17 years at time of surgery
* ACL full thickness lesion
* meniscal lesions repaired simultaneously
* completed research protocol

Exclusion Criteria:

* age <10 yo and >17 yo.
* PCL concomitant injury
* polytrauma
* other same knee surgeries performed before intervention

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Lachman test | up to six months
  Assessment of knee stability in sagittal plane (positive/negative)
Pivot shift test | up to six months
  Assessment of knee rotational stability (positive/negative)
Apley's distraction test | up to six months
  Assessment of knee rotational stability (positive/negative)
MRI evaluation | up to 12 months
  Assessment of reconstructed ACL morphology and degenerative changes of the knee - cartilage average volume (cubic centimeter) [cm3]
Isokinetic evaluation - peak torque | up to 12 months
  Quadriceps and hamstrings isokinetic tests in either 60 deg/s and 180 deg/s velocities with evaluation of peak torque (Newton-meter, [Nm])
Arthrometer testing | up to six months
  Assessment of knee stability in sagittal plane with digital arthrometer use (millimeters, [mm])
Isokinetic evaluation - torque at 30 deg | up to 12 months
  Quadriceps and hamstrings isokinetic tests in either 60 deg/s and 180 deg/s velocities with evaluation of torque at 30 deg (Newton-meter, [Nm])
Isokinetic evaluation - angle of peak torque | up to 12 months
  Quadriceps and hamstrings isokinetic tests in either 60 deg/s and 180 deg/s velocities with evaluation of angle of peak torque (degrees [deg]))
Isokinetic evaluation - time to peak torque | up to 12 months
  Quadriceps and hamstrings isokinetic tests in either 60 deg/s and 180 deg/s velocities with evaluation of time to peak torque (milliseconds [ms])
Isokinetic evaluation - work fatigue | up to 12 months
  Quadriceps and hamstrings isokinetic tests in either 60 deg/s and 180 deg/s velocities with evaluation of work fatigue (percent [%])

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Małecki, Ph.D., Study Director — Polish Mother Memorial Hospital Research Institute
Locations (1):
- Polish Mother Memorial Hospital Research Institute, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request via e-mail krzynormal@wp.pl
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2022-2028
Access Criteria: krzynormal@wp.pl